CLINICAL TRIAL: NCT01849094
Title: Evaluating the Safety, Pharmacokinetics and Haemodynamic Effect of a Slow Release Oral Formulation of Milrinone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Prof David Kaye, Head, Experimental Cardiology and Heart Failure Division Baker Heart Research Institute & Cardiologist, Heart Centre, Alfred Hospital, The Alfred
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DK-MIL-1
Record Dates: First submitted 2013-04-30; First posted 2013-05-08 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Healthy; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milrinone 6mg (Experimental): single oral dose of 6mg ER milrinone tablet (Part A).
  1. single intravenous infusion of milrinone (per Alfred Hospital protocol. 50ug/kg loading dose over 15 mins followed by infusion at 0.375 ug/kg/min for 6 hrs) - Part B.
  Interventions: Drug: milrinone 10mg ER; Drug: milrinone 14mg
- Milrinone 10mg ER (Active Comparator): single oral dose of 10 mg ER milrinone tablet (Part A) single oral dose of 10 mg ER milrinone tablet (Part B)
  Interventions: Drug: Milrinone 6mg; Drug: milrinone 14mg
- Milrinone 14mg (Active Comparator): single oral dose of 14 mg ER milrinone tablet (Part A) single dose of 14 mg ER milrinone tablet 4. single oral dose of 18 mg ER milrinone tablet (if the group average plasma milrinone levels is less than 150 ug/L with 15 mg dose) - (Part B)
  Interventions: Drug: Milrinone 6mg; Drug: milrinone 14mg

INTERVENTIONS:
Drug: Milrinone 6mg — Administration of study medications, PK sampling If Part B - add on 6 hour haemodynamic invasive measurements
  Arms: Milrinone 10mg ER; Milrinone 14mg
Drug: milrinone 10mg ER — Administration of study medications, PK sampling If Part B - add on 6 hour haemodynamic invasive measurements
  Other Names: Milirone
  Arms: Milrinone 6mg
Drug: milrinone 14mg — Administration of study medications, PK sampling If Part B - add on 6 hour haemodynamic invasive measurements
  Other Names: Milirone

SUMMARY:
To determine the pharmacokinetic profile of a new (extended release) formulation of milrinone and to demonstrate evidence of hemodynamic effect

Primary: Pharmacokinetic profile - to demonstrate stable plasma levels Secondary (HF cohort) - to demonstrate evidence of haemodynamic benefit

Study Design: Open label

ELIGIBILITY:
Inclusion Criteria:

* Part A: Healthy volunteers; Part B: Heart failure patients Inclusion Criteria - Part A Healthy Volunteers

Participants must:

1. Provide written informed consent prior to any study procedure and agree to adhere to all protocol requirements
2. Be aged between 18 to 45 years old inclusive at the time of consent
3. Be in good general health without clinically significant medical history
4. Have a body mass index (BMI) between 19- 30 kg/m2 inclusive
5. Documented 12-lead ECG with no clinically significant abnormalities, as determined by the Investigator
6. No clinically significant abnormalities in screening or Day 0 laboratory tests, as determined by the Investigator;
7. Female subjects of reproductive potential must have a negative serum pregnancy (β-HCG) test at screening and a negative urine pregnancy test at Day 0 prior to dosing. Female subjects must also be non-lactating
8. Negative Human Immunodeficiency Virus (HIV), Hepatitis B and Hepatitis C Screening test results

Inclusion Criteria - Part B Heart Failure Patients

Participants must:

1. Provide written informed consent prior to any study procedure and agree to adhere to all protocol requirements
2. Heart Failure patients with LVEF less than45%
3. NYHA II-III
4. Stable medications (for greater than 48hrs)
5. Systolic BP greater than 90

Exclusion Criteria:

* Exclusion Criteria - Part A Healthy Volunteers

Participants will not be enrolled if they meet any of the following criteria:

1. If female, pregnant or lactating
2. Receipt of any investigational agent or drug within 30 days or 5 half-lives (whichever is longer) prior to the first dose of Investigational product
3. Use of prescription drugs within 4 weeks prior to first dosing. Subjects who have used over the counter medication excluding paracetamol, topical over the counter medications and routine vitamins but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 7 days of first dosing, unless agreed as non-clinically relevant by the Principal Investigator
4. No clinically relevant findings in the medical history, laboratory examination and physical examination, especially with regards to cardiovascular system and renal function
5. A positive urine test for drugs of abuse or alcohol at Screening or on the day of admittance to the Study Unit
6. Normal dietary habits
7. Any major surgical procedure within one month of entry into the study
8. Have difficulties communicating reliably with the Investigator or unlikely to co-operate with the requirements of the study.
9. Any other condition which in the view of the Investigator is likely to interfere with study or put the subject at risk.

Exclusion Criteria - Part B Heart Failure Patients

1. Unstable heart failure including NYHA IV symptoms
2. Treatment with intravenous inotropes or mechanical circulatory support.
3. Unstable rhythm including frequent non-sustained ventricular tachycardia or poorly controlled atrial fibrillation (ventricular rate >100).
4. Severe renal impairment Cr>200umol/L or dialysis.
5. Life-threatening haematological, hepatic or pulmonary disease.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile - to demonstrate stable plasma levels | 0, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours
  Laboratory Analysis: Plasma milrinone concentration

SECONDARY OUTCOMES:
(Heart Failure cohort) - to demonstrate evidence of haemodynamic benefit | 6 hours
  ECG and Blood pressure and HR Monitoring Swan Ganz insertion for haemodynamic measurements (RA volume , RVSP, CO, PA, PAWP)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Alfred Hospital, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria